CLINICAL TRIAL: NCT02520999
Title: Comparison of the Effect of Various External Pressure on Blood During Rapid Infusion
Brief Title: The Effect of Various External Pressure on Blood
Acronym: EPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hyub Huh (Other)
Responsible Party: Sponsor-Investigator, Hyub Huh, M.D., Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BP300
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5days (Active Comparator): 5 days after blood sampling, various external pressure test will be done. Blood wil be stored in refrigerator(Celsius 4 degree) until study day. External pressure 0, 100, 150, 200, 250, 300mmHg will be applied to each blood sample.
  Interventions: Device: Auto PC(Acemedical, Goyang-si, Korea) - 0mmHg(control); Device: Auto PC(Acemedical, Goyang-si, Korea) - 150mmHg; Device: Auto PC(Acemedical, Goyang-si, Korea) - 200mmHg; Device: Auto PC(Acemedical, Goyang-si, Korea) - 250mmHg; Device: Auto PC(Acemedical, Goyang-si, Korea) - 300mmHg
- 35days (Active Comparator): 35 days after blood sampling, various external pressure test will be done. Blood wil be stored in refrigerator(Celsius 4 degree) until study day. External pressure 0, 100, 150, 200, 250, 300mmHg will be applied to each blood sample.
  Interventions: Device: Auto PC(Acemedical, Goyang-si, Korea) - 0mmHg(control); Device: Auto PC(Acemedical, Goyang-si, Korea) - 150mmHg; Device: Auto PC(Acemedical, Goyang-si, Korea) - 200mmHg; Device: Auto PC(Acemedical, Goyang-si, Korea) - 250mmHg; Device: Auto PC(Acemedical, Goyang-si, Korea) - 300mmHg

INTERVENTIONS:
Device: Auto PC(Acemedical, Goyang-si, Korea) - 0mmHg(control) — Blood pass through infusion set without external pressure.
Device: Auto PC(Acemedical, Goyang-si, Korea) - 150mmHg — Blood pass through infusion set under external pressure (150mmHg)
Device: Auto PC(Acemedical, Goyang-si, Korea) - 200mmHg — Blood pass through infusion set under external pressure (200mmHg)
Device: Auto PC(Acemedical, Goyang-si, Korea) - 250mmHg — Blood pass through infusion set under external pressure (250mmHg)
Device: Auto PC(Acemedical, Goyang-si, Korea) - 300mmHg — Blood pass through infusion set under external pressure (300mmHg)

SUMMARY:
Rapid infusion of blood is needed occasionally for control massive bleeding. For rapid infusion, external pressure can be used. The investigators will study correlation between external pressure and hemolysis and deformability of red blood cell.

DETAILED DESCRIPTION:
Rapid infusion of blood is needed occasionally for control massive bleeding. For rapid infusion, external pressure can be used which cause hemolysis and alteration of red blood cell. The investigators will study correlation between variable external pressure and hemolysis and deformability of red blood cell. Differ from previous study, the investigator will use scanning electron microscope for observation red blood cell.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers, without any underlying disease.

Exclusion Criteria:

* history of delivery, abortion in past 6 months.
* weight : male under 50kg, female under 45kg
* heart rate under 50 or over 100
* fever : over 37.5
* blood pressure : over 180/100

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Hemolysis and alteration of deformability of red blood cell caused by external pressure | 1hour

CONTACTS AND LOCATIONS:
Overall Officials: Hyub Huh, M.D., Study Director — Department of anesthesiology and pain medicine, Korea University Anam Hospital
Locations (1):
- Korea university anam hospital, Seoul, South Korea